CLINICAL TRIAL: NCT01066273
Title: Somatosensory Based Treatments for Tinnitus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator no longer at institution
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-12-056
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P-Stim device (Experimental): Receiving the device that is activated
  Interventions: Device: P-Stim

INTERVENTIONS:
Device: P-Stim — The P-Stim is a battery-powered, transcutaneous electrical stimulator that delivers 1 per second bipolar 1 millisecond pulses to three points on the auricle. The device connects via three fine insulated stainless steel wires to three needles (each 0.4 mm diameter, 2 mm long) that have been applied to three different points on the auricle. The device is powered by three zinc air batteries, each with a voltage of 1.4 V. The device is on for 180 minutes, then off for 180 minutes, for a maximum period of up to 96 hours. The battery and electronics are contained in a 6 mm by 2.5 mm pack that has one adhesive surface which is applied to the skin behind the ear. The adhesive is conductive and acts as the return for the device. The battery pack is secured with tape.

SUMMARY:
Studies have established that the somatosensory system of the upper cervical region and head can be intimately involved in tinnitus. Tinnitus can arise directly from a disorder of the head and upper neck via the somatosensory system. Our clinical experience and review of reports of various types of treatments support the hypothesis that treatment modalities involving the somatosensory system can benefit individuals whose tinnitus is likely on a somatosensory basis, namely people with symmetric hearing thresholds but asymmetric widely fluctuating tinnitus. However these previous studies did not (a) limit their treatment population to only people with tinnitus on a somatosensory basis and (b) did not assess their results by considering this tinnitus subpopulation separately from the entire group of tinnitus subjects they treated. Hence, the purpose of this study is to re-assess these treatments by targeting people whose audiograms can not account for their tinnitus, such as individuals with symmetric hearing thresholds but asymmetric widely fluctuating tinnitus

DETAILED DESCRIPTION:
Until recently our attempts over the years at treatment of patients with such types of tinnitus has met with little or no success. These treatments have included cervical physical therapy and dental treatments for bruxism. A few with such tinnitus responded have had some benefit from acupuncture applied to their periauricular region. A small formal trial with a few patients did not provide any relief.

However a literature review (Levine et al., 2007) found a consistent line of evidence for a tinnitus subgroup responsive to somatosensory based treatment modalities, including electrical stimulation in the periauricular region, and acupuncture. Furthermore an electrical stimulation device of the auricle P-Stim was found to be more effective than standard acupuncture for a variety of conditions, including chronic cervical and low back pain. For this convergence of reasons we have initiated an open trial with P-Stim over the past 11 months. In a sense we have used it in an "off-label" capacity; just as many medications have been found to be useful for conditions for which the medications were not developed (see Levine 2006).

The P-Stim is a battery-powered, transcutaneous electrical stimulator that delivers 1 per second bipolar 1 millisecond pulses to three points on the auricle. The device connects via three fine insulated stainless steel wires to three needles (each 0.4 mm diameter, 2 mm long) that have been applied to three different points on the auricle. The device is powered by three zinc air batteries, each with a voltage of 1.4 V. The device is on for 180 minutes, then off for 180 minutes, for a maximum period of up to 96 hours. The battery and electronics are contained in a 6 mm by 2.5 mm pack that has one adhesive surface which is applied to the skin behind the ear. The adhesive is conductive and acts as the return for the device. The battery pack is secured with tape.

We have met with some success using P-Stim for what appear to be two tinnitus subgroups: somatic pulsatile tinnitus syndrome (Levine et al., 2008) and patients with non-pulsatile unilateral fluctuating tinnitus associated with deep ear pain.

ELIGIBILITY:
Inclusion Criteria:

* Age range: above age 18

Exclusion Criteria:

* people with a bleeding disorder,
* and those on coumadin will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Quieter tinnitus | 6 months

IPD SHARING:
Plan to Share IPD: No